CLINICAL TRIAL: NCT00263731
Title: Preoperative Metabolomic Analysis of Primary Lung Cancer: A Translational Clinical Trial of the Brown Cancer Center
Brief Title: Metabolomic Analysis of Lung Cancer
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Donald Miller, Professor, University of Louisville
Other Study IDs: 523.05; BCC-LUN-05-002 (Other: James Graham Brown Cancer Center Clinical Trials Office)
Record Dates: First submitted 2005-12-07; First posted 2005-12-09 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Carcinoma, Non-Small Cell Lung; Carcinoma, Small Cell Lung
Keywords: lung cancer; non-small cell lung cancer; small cell lung cancer; cancer metabolism
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Lung Neoplasms | interventions — 1,2-O-isopropylidene-D-glucofuranose

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group 1 (Experimental Group): 250 subjects with suspected or confirmed lung cancer undergoing surgical resection, will receive 13-C-glucose prior to surgery
  Interventions: Other: 13-C-glucose
- Group 2 (Control Group): 250 subjects with suspected or confirmed lung cancer undergoing surgical resection, will not receive 13-C-glucose prior to surgery
- Group 3 (Healthy Subjects): 250 healthy subjects (must be at least 30 years of age and have no prior history of diagnosed lung cancer) will provide 1 blood sample and 1 urine sample.

INTERVENTIONS:
Other: 13-C-glucose — 10 grams of 13-C-glucose intravenously, as a 30-minute "piggyback" infusion, 2 to 6 hours prior to scheduled surgical resection of primary lung cancer.
  Groups: Group 1 (Experimental Group)

SUMMARY:
The purpose of this study is to learn more about the metabolic properties of lung cancer cells.

DETAILED DESCRIPTION:
It has long been known that cancer cells absorb and break down substances in the body differently than healthy, non-cancer cells. This process of absorbing and breaking down substances is known as metabolism and is increased in cancer cells. Recent research suggests that this increased metabolic activity makes it easier for cancer cells to multiply. The objective of the study is to characterize the metabolism of glucose by lung tumors by serum metabolite analysis, using a variant of glucose (sugar) which makes up 1% of glucose in nature.

ELIGIBILITY:
Lung Cancer Patients (Groups 1 & 2)

Inclusion Criteria:

* patients with suspected, clinically diagnosed, or histologically diagnosed lung cancer. Occasionally, other cancers (including metastatic cancers to the lung) may be resected for the study as negative controls for NSCLC, as warranted by the particulars of the case.
* patients must have general medical conditions to allow them to undergo surgical resection of their primary tumor

Exclusion Criteria:

* history of diabetes for the experimental group (surgery + glucose); patients with a history of diabetes are allowed in the control group (surgery/no glucose)
* known hepatitis C or HIV (AIDS)

Healthy Subjects (Group 3)

Inclusion Criteria:

* at least 30 years of age
* preferably be fasting for 12 hours (minimum 8 hours) prior to enrollment

Exclusion Criteria:

* prior history of diagnosed lung cancer
* known hepatitis C or HIV (AIDS)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Group 1 (experimental group): 250 lung cancer patients undergoing surgery, with 13-C-glucose infusion);
  * Group 2 (control group): 250 lung cancer patients undergoing surgery, without 13-C-glucose infusion); and
  * Group 3 (healthy subjects): 250 subjects to provide 1 blood sample and 1 urine sample.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2005-12; Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
metabolic profiles of cancerous vs. healthy lung tissue | after 13-C-glucose infusion

SECONDARY OUTCOMES:
glycolytic metabolism in plasma | before and after 13-C-glucose infusion
metabolic markers in urine | collected during surgery
metabolic markers in serum | before and after 13-C-glucose infusion
metabolic markers in bronchoalveolar fluid | during diagnostic bronchoscopy or during surgery
metabolic markers in expired breath | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Donald M Miller, MD, PhD, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, University of Louisville, Louisville, Kentucky, United States

REFERENCES:
- See also: James Graham Brown Cancer Center — http://www.browncancercenter.org